CLINICAL TRIAL: NCT07177872
Title: A Multicenter, Open-label Study Evaluating the Long-term Efficacy and Safety of NTQ5082 Capsules in the Treatment of Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Long-term Efficacy and Safety of NTQ5082 Capsules
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTQ5082-PNH-302
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTQ5082 (Experimental): NTQ5082
  Interventions: Drug: NTQ5082 capsules 200 mg

INTERVENTIONS:
Drug: NTQ5082 capsules 200 mg — NTQ5082 capsules 200 mg

SUMMARY:
NTQ5082 capsules are a small molecule CFB inhibitor. This study is a multicenter, open-label study evaluating the long-term efficacy and safety of NTQ5082 capsules in the treatment of patients with paroxysmal nocturnal hemoglobinuria

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥ 18 years, regardless of gender. 2) Subjects who have previously received and completed NTQ5082 study treatment and, as determined by the investigator, have benefited from treatment and are likely to benefit from continued NTQ5082 treatment, or subjects in the control group receiving eculizumab.

  3) Subjects who have received ACYW135 group meningococcal and pneumococcal vaccines as required by the previous protocol, and whose vaccine protection period, as determined by the investigator, falls within the treatment duration of this study.

  4) Subjects who agree to use at least one effective contraceptive method during sexual intercourse with their partner from the time they sign the informed consent form until 4 weeks after the last dose, refrain from cryopreservation of sperm or eggs, and refrain from sperm or egg donation.

  5) Subjects who agree to sign the informed consent form and commit to abide by all study regulations.

Exclusion Criteria:

* 1) Previous history of bone marrow/hematopoietic stem cell or solid organ transplant (e.g., heart, lung, kidney, liver).

  2) Previous history of splenectomy. 3) Previous history of recurrent invasive infection with encapsulated bacteria (e.g., meningococci, Streptococcus pneumoniae), previous history of systemic anti-tuberculosis treatment, or current tuberculosis infection.

  4) History of malignancy within 5 years prior to screening, excluding cured localized basal cell carcinoma of the skin, squamous cell carcinoma of the skin, papillary thyroid carcinoma, or carcinoma in situ of the cervix.

  5) Known or suspected hereditary complement deficiency or primary or severe secondary immunodeficiency. 6) Patients with a history of clinically significant kidney, heart, liver, or lung disease who are deemed unsuitable for participation by the investigator, including but not limited to severe kidney disease (e.g., eGFR <30 mL/min/1.73 m²), advanced heart disease (e.g., NYHA class IV), or severe lung disease (e.g., severe pulmonary hypertension (WHO class IV).

  7) Patients suspected of being allergic to the study drug or any component of the study drug.

  8) Pregnant or lactating female subjects. 9) Other conditions deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 96 Weeks

SECONDARY OUTCOMES:
the proportion of subjects with hemoglobin (HB) levels ≥ 120 g/L without red blood cell (RBC) transfusion | 96 weeks
the change in hemoglobin level compared to before NTQ5082 capsule treatment without red blood cell transfusion | 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences ,, Tianjin, Tianjin Municipality, China